CLINICAL TRIAL: NCT04132232
Title: Smoking Reduction In Gravid Women With Substance Use Disorders (SIGS): A Randomized Controlled Trial
Brief Title: Smoking Reduction In Gravid Substance Use Disorders
Acronym: SIGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rubymel J Knupp, Maternal-Fetal Medicine Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIGS; JCHF (Other Grant/Funding Number: Jefferson County Health Fund); UAB (Other Grant/Funding Number: University of Alabama Ob/Gyn Fund for Excellence in Education)
Record Dates: First submitted 2019-10-12; First posted 2019-10-18 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Smoking in Mother Complicating Pregnancy; Tobacco Use Disorder; Tobacco Smoking
Keywords: smoking in pregnancy; substance use disorder; carbon monoxide; fetal carboxyhemoglobin
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Will not discuss percent fetal carboxyhemoglobin to control group versus disclosing percent fetal carboxyhemoglobin to intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): 1. The patient will exhaled into the Smokerlyzer® device will at each visit
  2. Exhaled carbon monoxide and fetal carboxyhemoglobin levels will be disclosed to the patient
  3. Risks of adverse perinatal outcomes related to maternal carboxyhemoglobin and fetal carboxyhemoglobin level will be provided.
  Interventions: Diagnostic Test: knowledge of expired maternal carbon monoxide and fetal carboxyhemoglobin levels
- Control Group (No Intervention): 1. The patient will exhale into the Smokerlyzer® device at each visit.
  2. Exhaled carbon monoxide and fetal carboxyhemoglobin level will NOT be disclosed to the patient
  3. No risks of adverse perinatal outcomes related to maternal carbon monoxide and fetal carboxyhemoglobin levels will be provided

INTERVENTIONS:
Diagnostic Test: knowledge of expired maternal carbon monoxide and fetal carboxyhemoglobin levels — Will use the Smokerlyzer® device at each visit and be provided information on exhaled carbon monoxide and fetal carboxyhemoglobin. Risks of adverse perinatal outcomes related to maternal carbon monoxide and fetal carboxyhemoglobin level will be provided.
  Other Names: adverse outcomes related to expired maternal carbon monoxide and fetal carboxyhemoglobin levels
  Arms: Treatment Group

SUMMARY:
The aim of this study is to encourage smoking cessation in women with substance use disorders by providing knowledge of expired carbon monoxide. We hypothesize that women who are provided knowledge of their expired carbon monoxide and the associated percent fetal carboxyhemoglobin will have a greater success at quitting smoking during pregnancy than women who are not provided this information.

A secondary aim of the study is to correlate expired carbon monoxide throughout pregnancy with infant birth weight.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Pregnant smokers who are substances users who meet inclusion criteria will be offered participation in the study at their first obstetrical appointment. Patients who consent to participate will be randomized.

At the enrollment/randomization visit, women will be randomized to either the intervention (knowledge of and interpretation carbon monoxide levels and associated percent fetal carboxyhemoglobin) or control group (no information on carbon monoxide and associated percent fetal carboxyhemoglobin). Allocation will be computer generated. This will be done after the patient meets all inclusion criteria. If randomization to the intervention arm, the patient will be notified of carbon monoxide and associated fetal carboxyhemoglobin levels at each obstetrical visit and counseled on how it affects maternal and fetal health.

If randomized to the control arm, the patient will have expired carbon monoxide and associated fetal carboxyhemoglobin levels measured at each obstetrical visit but blinded to these results. These patients will not be notified of the levels, nor counseled on what levels mean for maternal or fetal health.

See below for intervention and control protocols.

Maternal demographic (age, race, socioeconomic status), medical history (other medical problems, medications, height, weight) and obstetric history (parity, gestational age) data will be abstracted from the patient's chart and supplemented with a patient questionnaire at the enrollment/randomization visit. The primary outcome is the expired maternal carbon monoxide level at the last obstetric visit or at delivery. This will be determined by the Smokerlyzer device used to measure this. Secondary aims of the study will be to evaluate how maternal carbon monoxide levels correlate with fetal growth, cigarette use per day, patient satisfaction and neonatal birth weight.

All patients will have the following performed at the enrollment/randomization visit and subsequent prenatal visits:

a. The order of events for all patients will be as follows: i. Blood pressure evaluation ii. Weight iii. Fundal height iv. Patient will be asked the number of cigarettes used per day v. Patient will exhale into Smokerlyzer device to obtain expired carbon monoxide and associated percent fetal carboxyhemoglobin vi. Patients will be provided smoking cessation resources and counseling on smoking cessation in pregnancy

Intervention Protocol

1. Intervention group will undergo Smokerlyzer ® exhaled carbon monoxide measurements at enrollment, each prenatal visit, and at their last (>36 week) prenatal visit or at delivery if not captured in clinic.
2. Women will be informed of their exhaled carbon monoxide measurement at each visit as well as the correlation to fetal carboxyhemoglobin.
3. At each visit, the intervention group will receive counseling on fetal impact of smoking based on fetal carboxyhemoglobin level and institutional and state information on smoking cessation will be provided.
4. The patient will then proceed to the remainder of the obstetrical visit.

Control Protocol

1. Women in the control group will undergo Smokerlyzer ® exhaled carbon monoxide measurements at enrollment, each prenatal visit and at their final (>36 week) prenatal visit or at delivery if not captured in clinic.
2. Both levels (maternal carbon monoxide and fetal carboxyhemoglobin) will be recorded by the co-investigatory, but NOT disclosed to the patient
3. At each visit, control group will be provided institutional and state information on smoking cessation if they report continued smoking.
4. The patient will then proceed to remainder of the obstetrical visit.

For both groups:

At the time of delivery, maternal and neonatal outcome data will be recorded from the chart, including gestational age at delivery, mode of delivery, indications for delivery, birth weight, Apgar score, cord blood gas, length of stay, and neonatal complications, if any. A survey will be completed for both intervention and standard care groups after delivery.

ELIGIBILITY:
Inclusion Criteria:

i. Age 16-45

ii. Singleton gestation

iii. Gestational age at enrollment <24 weeks

iv. Substance use disorder defined as modified National Institute on Drug Abuse ASSIST ≥4

v. Cigarette smoker using ≥10 cigarettes/day interested in quitting

Exclusion criteria:

i. Known or suspected fetal growth restriction at enrollment

ii. Known fetal anomaly, aneuploidy, or demise

iii. Not interested in smoking cessation or reduction during pregnancy

iv. E-cigarette use

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women and neonates: male and females
Enrollment: 74 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel G Sinkey, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandberg A, Skold CM, Grunewald J, Eklund A, Wheelock AM. Assessing recent smoking status by measuring exhaled carbon monoxide levels. PLoS One. 2011;6(12):e28864. doi: 10.1371/journal.pone.0028864. Epub 2011 Dec 16. PMID 22194931
- [Background] Bedfont. Smokerlyzer range user manual. http://www.bedfont.com/file.php?f=ZmlsZSMjMTgxMg. Updated 2019. Accessed Sept 16, 2016.
- [Background] Gomez C, Berlin I, Marquis P, Delcroix M. Expired air carbon monoxide concentration in mothers and their spouses above 5 ppm is associated with decreased fetal growth. Prev Med. 2005 Jan;40(1):10-5. doi: 10.1016/j.ypmed.2004.04.049. PMID 15530575
- [Background] Goldstein AO, Gans SP, Ripley-Moffitt C, Kotsen C, Bars M. Use of Expired Air Carbon Monoxide Testing in Clinical Tobacco Treatment Settings. Chest. 2018 Feb;153(2):554-562. doi: 10.1016/j.chest.2017.11.002. Epub 2017 Nov 11. PMID 29137909
- [Background] Riaz M, Lewis S, Coleman T, Aveyard P, West R, Naughton F, Ussher M. Which measures of cigarette dependence are predictors of smoking cessation during pregnancy? Analysis of data from a randomized controlled trial. Addiction. 2016 Sep;111(9):1656-65. doi: 10.1111/add.13395. Epub 2016 May 6. PMID 26997495
- [Background] Jha P, Ramasundarahettige C, Landsman V, Rostron B, Thun M, Anderson RN, McAfee T, Peto R. 21st-century hazards of smoking and benefits of cessation in the United States. N Engl J Med. 2013 Jan 24;368(4):341-50. doi: 10.1056/NEJMsa1211128. PMID 23343063
- [Background] QuickStats: Number of Deaths from 10 Leading Causes,* by Sex - National Vital Statistics System, United States, 2015. MMWR Morb Mortal Wkly Rep. 2017 Apr 21;66(15):413. doi: 10.15585/mmwr.mm6615a8. PMID 28426642
- [Background] Middleton ET, Morice AH. Breath carbon monoxide as an indication of smoking habit. Chest. 2000 Mar;117(3):758-63. doi: 10.1378/chest.117.3.758. PMID 10713003
- [Background] McClure JB. Are biomarkers a useful aid in smoking cessation? A review and analysis of the literature. Behav Med. 2001 Spring;27(1):37-47. doi: 10.1080/08964280109595770. PMID 11575171
- [Background] 11. Bedfont. Smokerlyzer range user manual. http://www.bedfont.com/file.php?f=ZmlsZSMjMTgxMg. Updated 2019. Accessed Sept 16, 2019.
- [Background] Shahab L, West R, McNeill A. A randomized, controlled trial of adding expired carbon monoxide feedback to brief stop smoking advice: evaluation of cognitive and behavioral effects. Health Psychol. 2011 Jan;30(1):49-57. doi: 10.1037/a0021821. PMID 21299294
- [Background] Bize R, Burnand B, Mueller Y, Rege-Walther M, Camain JY, Cornuz J. Biomedical risk assessment as an aid for smoking cessation. Cochrane Database Syst Rev. 2012 Dec 12;12:CD004705. doi: 10.1002/14651858.CD004705.pub4. PMID 23235615
- [Background] Reynolds CME, Egan B, Kennedy RA, O'Malley E, Sheehan SR, Turner MJ. The implications of high carbon monoxide levels in early pregnancy for neonatal outcomes. Eur J Obstet Gynecol Reprod Biol. 2019 Feb;233:6-11. doi: 10.1016/j.ejogrb.2018.11.020. Epub 2018 Nov 30. PMID 30529257
- [Background] Ecker J, Abuhamad A, Hill W, Bailit J, Bateman BT, Berghella V, Blake-Lamb T, Guille C, Landau R, Minkoff H, Prabhu M, Rosenthal E, Terplan M, Wright TE, Yonkers KA. Substance use disorders in pregnancy: clinical, ethical, and research imperatives of the opioid epidemic: a report of a joint workshop of the Society for Maternal-Fetal Medicine, American College of Obstetricians and Gynecologists, and American Society of Addiction Medicine. Am J Obstet Gynecol. 2019 Jul;221(1):B5-B28. doi: 10.1016/j.ajog.2019.03.022. Epub 2019 Mar 27. No abstract available. PMID 30928567
- See also: Smokerlyzer product website — https://www.covita.net/product/microbaby-smokerlyzer/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: 1. The patient will exhaled into the Smokerlyzer® device will at each visit
  2. Exhaled carbon monoxide and fetal carboxyhemoglobin levels will be disclosed to the patient
  3. Risks of adverse perinatal outcomes related to maternal carboxyhemoglobin and fetal carboxyhemoglobin level will be provided.
  knowledge of expired maternal carbon monoxide and fetal carboxyhemoglobin levels: Will use the Smokerlyzer® device at each visit and be provided information on exhaled carbon monoxide and fetal carboxyhemoglobin. Risks of adverse perinatal outcomes related to maternal carbon monoxide and fetal carboxyhemoglobin level will be provided.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 37 | 37
Completed | 30 | 29
Not Completed | 7 | 8
Not completed — Randomized but met exclusion criteria. | 1 | 1
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (6.9) | 32.4 (9.4) | 31.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 26 | 24 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Expired Maternal Carbon Monoxide Level at randomization [Mean (Standard Deviation); unit: ppm] | 15.4 (8.8) | 11.2 (5.5) | 13.4 (7.6)
Average number of cigarettes per day at enrollment [Mean (Standard Deviation); unit: cigarettes] | 12.3 (3.8) | 12.6 (4.4) | 12.4 (4.09)

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Smoking ≥ 10 Cigarettes/Day in Each Group at Final Measurement by Exhaled Carbon Monoxide Level
Description: Prevalence of smoking ≥ 10 cigarettes/day in each group at final measurement by exhaled carbon monoxide level at last prenatal visit prior to delivery, as measured by exhaled carbon monoxide
Time Frame: Final measurement (last prenatal care visit or at delivery)
Population: Participants who had expired carbon monoxide measured at either their last prenatal visit or at delivery.
Measure: Number; unit: participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 37 | 36
participants | 22 | 16
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.06, Chi-squared

ADVERSE EVENTS:
Time Frame: Over the course of the study period, which is around 10 months per participant.
Description: As this is a low-risk study, an independent data safety monitoring board will not be formed.
  We defined an adverse event as an undesirable experience or outcome occurring in a research participant, regardless of whether participation in the research study caused the event to occur. For example, placental abruption and/or stillbirth are known risks of pregnancy, and while not associated with the Smokerlyzer® device, would be considered an adverse event if it occurred during the study.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04132232/Prot_SAP_ICF_000.pdf